CLINICAL TRIAL: NCT06812585
Title: The Effect of Metformin As an Adjuvant Therapy on Immunological Parameters in Egyptian Patients with RRMS: a Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German University in Cairo (Other)
Responsible Party: Principal Investigator, Mohamed Youssef Elsayed, The Effect of Metformin as an Adjuvant Therapy on Immunological Parameters in Egyptian Patients with RRMS: A Pilot Study, German University in Cairo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MET in sNFL and NFK-B
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2022-04

CONDITIONS: Multiple Sclerosis (MS) - Relapsing-remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Active Comparator: Interferon beta 1 a (Rebiff ® 44mcg or Avonex ®) Interferon beta 1 a (Rebiff ® 44mcg or Avonex ®)
  Interventions: Other: Usual Care
- Intervention group (Experimental): Experimental: Metformin (Cidophage®) and Interferon Beta 1 a (Rebiff ® 44mcg or Avonex ®) Metformin 1000 mg (Cidophage® 1000 mg tablets, CID, Giza, Egypt) tablet twice daily for 6 months as add on therapy with Interferon beta 1 a (Rebiff ® 44mcg or Avonex ®).
  Interventions: Drug: Metformin (Cidophage®)

INTERVENTIONS:
Drug: Metformin (Cidophage®) — Antidiabetic agent used to treat type 2 diabetes, and to prevent type 2 diabetes.
  Arms: Intervention group
Other: Usual Care — Active Comparator: Interferon beta 1 a (Rebiff ® 44mcg or Avonex ®) Interferon beta 1 a (Rebiff ® 44mcg or Avonex ®)
  Arms: Control group

SUMMARY:
This pilot study aims to investigate the tolerability and feasibility of using metformin as an adjuvant treatment for RRMS. Also, it aims to evaluate the preliminary evidence of its efficacy by analyzing outcomes related to immunology, clinical manifestations, and radiological findings.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18 and 50 years of age who met the 2017 McDonald criteria were recruited.
* Patients with RRMS and had an EDSS score below 7.0.
* Participants were required to have been on a stable IFNβ-1a regimen for at least six months before the commencement of the study.

Exclusion Criteria:

* Individuals taking metformin or other diabetes medications, pregnant, and breastfeeding females were excluded.
* Those with congestive heart failure, liver impairment, kidney dysfunction, or chronic respiratory conditions were not eligible to participate.
* Additionally, patients who had undergone corticosteroids before or within 4 weeks of the study's commencement were ineligible for participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Change in serum levels of neurofilament light chain in both arms | After 6 months

SECONDARY OUTCOMES:
Change in serum levels of nuclear factor kappa B in both arms | After 6 months
Degree of remyelination visualized by MRI, it depends on clinician's overview. | After 6 months
Degree of disability assessed by Expanded Disability Status Scale. | After 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nasser Institute for Research and Treatment, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdelgaied MY, Abdelgawad O, Rashad MH, Solayman MH, El-Tayebi HM. Efficacy and tolerability of metformin as an adjuvant therapy in patients with relapse-remitting multiple sclerosis receiving interferon Beta 1a: A randomized pilot trial. J Neuroimmunol. 2026 Mar;412:578852. doi: 10.1016/j.jneuroim.2025.578852. Epub 2025 Dec 31. PMID 41483718